CLINICAL TRIAL: NCT04863833
Title: Diagnostic Value of Digital Breast Tomosymthesis for Breast Mass Lesions Characterization
Brief Title: Tomosymthesis for Breast Mass Lesion Characterization
Acronym: DBT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Asmaa Abdelmonem Ahmed (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Asmaa Abdelmonem Ahmed, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Tomosymthesis
Record Dates: First submitted 2021-03-06; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Female Breast Cancer
Keywords: Tomosyntheses, X-ray--Digital Tomosynthesis-- Breast Tomosyntheses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
To Estimate diagnostic value of tomo synthesis for breast mass lesions characterization ( shape, margin, and density, detail of mass margins, Differences in mass density , Tumor measurement,.)

DETAILED DESCRIPTION:
Breast lesions are observed in about 20% of female patients1. However this percentage is likely to represent an underestimation of the true incidence of these lesions because breast imaging (MRI, ultrasound or mammography) was performed in only a small number of the patients of these series. The lesions are possibly palpable and most of the time asymptomatic2.

In current clinical practice, mammography is the standard imaging modality for breast cancer screening and diagnosis.3 The advantages of mammography include a reasonably high sensitivity, high resolution, and low patient dose. However, a mammogram still suffers from being a two-dimensional projection of a three-dimensional object. The resulting overlap of normal fibro glandular tissue cannot only obscure the detection and characterization of lesions but also present false alarms leading to unnecessary recall studies.4-6 To address this key limitation of mammography, 3D x-ray imaging techniques have been developed, including dedicated breast computed tomography (CT), which takes cone-beam x-ray projection images of the uncompressed breast in a full 360° scan, thus enabling reconstruction of a 3D breast volume 6-10 Digital x-ray tomosynthesis11,12(often abbreviated as "tomo") for the breast is a form of limited-angle cone-beam CT.13-14 A restricted number of projection images are acquired in an arc in the conventional mammography projection geometry, while the breast is compressed adjacent to the detector. Although some information is lost due to angular under sampling, breast tomo still creates a 3D volume at a dose comparable to that of traditional mammography. Moreover, the tomo device itself is usually based on an existing full-field digital mammography (FFDM) system. Although compression is required, this ensures proper posterior tissue coverage, immobilization to minimize motion artifacts, and a low dose.15The similarity of tomo to FFDM in terms of patient positioning, image acquisition, and aspects of image display suggests that there is minimal retraining required for the technologist or radiologist.16 As such, breast tomo synthesis is a 3D breast imaging modality with the potential to replace mammography17

. DBT offers potential advantages for evaluating masses, areas of architectural distortion, and asymmetries compared with those of conventional 2D mammographic images 18 In diagnostic settings, DBT improves work-up efficiency and the selection of patients recommended for biopsy, thereby reducing associated costs and additional imaging studies including additional mammographic views and unnecessary biopsies 19

ELIGIBILITY:
Inclusion Criteria:

female patients who undergoes DBT must have a compressed breast thickness of more than 2 cm,with small mass,age>35,not have mastitis,not proceed breast implant

Exclusion Criteria:

* Female Patients with breast implant ,severe nipple discharge, large palpable mass, mastitis and women within reproductive age(15-35 ) Female patients with huge breast that may exceed the detector size requirements for global diagnostic DBT.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self representative of gender identity
Study Population: All female patients except mentioned in exclusion criteria
  . Female patients who undergoes DBT must have a compressed breast thickness of more than 2 cm; therefore, some patients will not qualify
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
diagnosis of breast mass lesions | 2 years
  Mass regular in shape or not, homogeneous in echogenicity or not,calicfied or not,has speculation or not,single or multiple

SECONDARY OUTCOMES:
characters of benign and malignant breast mass | 2 years
  Mass invasive to all breast layer or not ,sarcoma,carcinoma or lymphoma,lymph node metastasis or not, secondary metastasis or not ,staging byTNM score, treatment by radical mastectomy or conservative mastectomy, distracted shape of breast or not